CLINICAL TRIAL: NCT01538381
Title: Neoadjuvant Afatinib Based Treatment Strategies Followed by Surgery in Squamous Cell Carcinoma of the Head and Neck: an EORTC NOCI-HNCG Window Study.
Brief Title: Neoadjuvant Afatinib Window Study in Squamous Cell Carcinoma of the Head and Neck
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Collaborators: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EORTC-90111-24111; 2011-005820-17 (EudraCT Number)
Record Dates: First submitted 2012-02-20; First posted 2012-02-24 (Estimated); Last update posted 2018-07-09 (Actual); Status verified 2018-07

CONDITIONS: Carcinoma, Squamous Cell of Head and Neck
Keywords: Neoadjuvant targeted therapy; Preoperative targeted therapy; Afatinib
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Afatinib; Observation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Afatinib (Experimental): Afatinib given orally for 2 weeks after randomization till day -1 prior to surgery (day 0) at a dose of 40 mg/day
  Interventions: Drug: Afatinib
- Observation (Other): No treatment only observation
  Interventions: Other: Observation

INTERVENTIONS:
Drug: Afatinib — Afatinib for 2 weeks at a dose of 40 mg/day
  Arms: Afatinib
Other: Observation — Observation
  Arms: Observation

SUMMARY:
The general objectives are to evaluate the pre-operative activity and the safety of afatinib in head and neck cancer and to explore the different downstream molecular pathways to identify tumor response and resistance mechanisms. The results from this study can be used to conduct a larger trial that would allow us to confirm or validate the hypotheses generated.

DETAILED DESCRIPTION:
This is a randomized, multicenter early phase II trial exploring the pre-operative activity of afatinib vs. nontreatment. The study includes an early monitoring of the surgical co-morbidities for patients treated with afatinib and accrual may be stopped prematurely according to a pre-defined safety stopping rule.

Patients will be randomized with a 5:1 ratio, between the two arms: afatinib and 'no treatment'. It is intended to include a total of 30 eligible patients out of which 25 patients will be randomized into the afatinib arm.

Patients allocated to the 'no treatment' arm will mainly serve as a reference to interpret the results of the translational research part of the study although no formal comparison between the afatinib arm and the 'no treatment' arm is intended.

Patients will be first registered into the EORTC system after signing the informed consent form. The site will have to complete all the study related procedures within 4 weeks prior randomization and all eligibility criteria should be met before the patient can be randomized into the study.

The registration of patients will proceed with slots for patients which will be opened or closed based on the randomization of patients into the afatinib arm. Starting with 3 free slots, an additional slot will become available for each patient randomized to the 'no treatment' arm.

Registration will be paused after three completes the 4 week observation period after surgery. Similar action will be done after the next 3 patients have been entered into the afatinib arm.

Once the first 6 patients in the afatinib arm have been observed for surgical toxicities of grade ≥ 3 for 4 weeks following surgery, the slot system will cease to operate.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed histologically proven squamous cell carcinoma of the oral cavity, oropharynx, hypopharynx or larynx.
* Patients selected for a primary surgical treatment
* Age ≥18 years
* Performance status ECOG 0-1
* Within 2 weeks prior randomization:

  * Adequate bone marrow function as demonstrated by neutrophils count ≥ 1,500/mm3, platelet count ≥ 75,000/mm3, WBC ≥ 3.0/109 L
  * Adequate hepatic function as demonstrated by bilirubin < 2 times upper limit of normal (ULN), ALAT or ASAT < 3 times ULN
  * Adequate renal function as demonstrated by serum creatinine <or= 1.5 mg/dL (< 133 µmol/L) or calculated creatinine clearance ≥50 mL/min
  * Controlled blood pressure (<140/90 mm Hg) with or without antihypertensive treatment
  * Prothrombin time (PT) with an international normalized ratio (INR) <or=1.2
  * Partial thromboplastin time (PTT) <or= 1.2 times ULN
  * Adequate cardiac function assessed by 12-lead ECG and if clinically indicated echocardiography to document LVEF
  * FDG-PET/CT performed
  * DCE MRI and DWI MRI performed
* Primary tumor ≥2 cm in their largest diameter measured bidimensionally by imaging done within 2 weeks prior to randomization
* Availability of tumor and normal mucosa biopsies during staging endoscopy (please refer to surgical guidelines for further information).
* Availability of blood samples for translational research
* Absence of any serious underlying medical conditions which could impair the ability of the patient to participate in the study
* Women of childbearing potential (WOCBP) must be using an adequate method of contraception to avoid pregnancy throughout the study and 6 months beyond stop of treatment in such a manner that the risk of pregnancy is minimized. In general, the decision for appropriate methods to prevent pregnancy should be determined by discussions between the investigator and the study subject. WOCBP include any female who has experienced menarche and who has not undergone successful surgical sterilization (hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or is not postmenopausal. Females should not be breast feeding.

  * Post menopause is defined as: amenorrhea ≥ 12 consecutive months without another cause or for women with irregular menstrual periods and on hormone replacement therapy (HRT), a documented serum follicle stimulating hormone (FSH) level > 35 mIU/mL
  * Women who are using oral contraceptives, other hormonal contraceptives (vaginal products, skin patches, or implanted or injectable products), or mechanical products such as an intrauterine device or barrier methods (diaphragm, condoms, spermicide) to prevent pregnancy, or are practicing abstinence or where their partner is sterile (e.g., vasectomy) should be considered to be of childbearing potential.
  * Women of child bearing potential must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 72 hours prior to the start of investigational product.
  * Female patients within one year of entering the menopause must agree to use an effective non-hormonal method of contraception during the treatment period and for at least 6 months after the last study treatment.
* Males must agree to use an effective method of contraception during the treatment period and for at least 6 months after the last study treatment.
* Absence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before registration in the trial
* Before patient registration, written informed consent must be given according to ICH/GCP, and national/local regulations

Exclusion Criteria:

* Patients with nasopharynx, nasal cavity and paranasal sinuses carcinomas, or recurrent/metastatic SCCHN are not eligible for this study
* T3 -T4 hypopharyngeal SCCHN are excluded.
* Distant metastases
* Active second malignancy during the last five years except non melanomatous skin cancer or carcinoma in situ of the cervix
* Prior chemotherapy, radiotherapy or targeted therapy including HER inhibitors (monoclonal antibodies or tyrosine kinase inhibitors) for SCCHN
* Concomitant use of potent P-gp inhibitors, potent P-gp inducers or Erythropoietin (EPO)
* Evidence of diabetes
* Evidence of interstitial lung disease
* Weight loss of more than 10% in the previous 6 months
* Participation in another interventional clinical trial in the preceding 30 days prior to randomization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2012-07; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Reduction of tumor Standardised Uptake Volume as assessed by FDGPET | Baseline and after two weeks of treatment
  Afatinib will be given orally for 2 weeks from the day of randomization until day -1 prior to surgery at a dose of 40 mg/day.Pre-treatment biopsies and blood samples will be harvested during the regular diagnosis staging procedure and at surgery.FDG-PET/CT-scan and MRIs will be performed before treatment (before day -15) and the day before surgery.The primary outcome measure is the reduction in the tumor standardised uptake volume as assessed by FDGPET

SECONDARY OUTCOMES:
Evaluation of tumour response to treatment by different imaging modalities like DWIMRI and DCEMRI | Baseline and after two weeks of treatment
  Response after 2 weeks of treatment, prior to surgery, evaluated by:
  * RECIST v1.1 using conventional imaging
  * Dynamic Contrast Enhanced Magnetic Resonance Imaging (DCE MRI)
  * Diffusion Weighted Imaging Magnetic Resonance Imaging (DWI MRI)

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Pascal Machiels, MD, Study Chair — European Organisation for Research and Treatment of Cancer - EORTC; Lisa Licitra, MD, Principal Investigator — European Organisation for Research and Treatment of Cancer - EORTC
Locations (4):
- Belgium (3):
  - Institut Jules Bordet, Brussels
  - Cliniques Universitaires St. Luc, Brussels
  - U.Z. Leuven - Campus Gasthuisberg, Leuven
- Istituto Nazionale Per Lo Studio E La Cura Dei Tumori, Milan, Italy

REFERENCES:
- [Derived] Machiels JP, Bossi P, Menis J, Lia M, Fortpied C, Liu Y, Lhommel R, Lemort M, Schmitz S, Canevari S, De Cecco L, Guzzo M, Bianchi R, Quattrone P, Crippa F, Duprez T, Lalami Y, Quiriny M, de Saint Aubain N, Clement PM, Coropciuc R, Hauben E, Licitra LF. Activity and safety of afatinib in a window preoperative EORTC study in patients with squamous cell carcinoma of the head and neck (SCCHN). Ann Oncol. 2018 Apr 1;29(4):985-991. doi: 10.1093/annonc/mdy013. PMID 29346507